CLINICAL TRIAL: NCT02931578
Title: Glycemic Index of Commonly Consumed Sweeteners
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI unexpectedly passed away, study future to be determined
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1604017520
Record Dates: First submitted 2016-10-07; First posted 2016-10-13 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Healthy
Keywords: glycemic index
MeSH Terms: interventions — Glucose Tolerance Test

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Glucose100 (Active Comparator): Participants in this arm will randomly receive 100% glucose in the OGTT drink 3 out of 9 visits.
  Interventions: Other: Glucose100; Other: Oral Glucose Tolerance Test
- Glucose50 (Active Comparator): Participants in this arm will randomly receive 50% glucose in the OGTT drink 3 out of 9 visits.
  Interventions: Other: Glucose50; Other: Oral Glucose Tolerance Test
- Glucose42 (Active Comparator): Participants in this arm will randomly receive 42% glucose in the OGTT drink 3 out of 9 visits.
  Interventions: Other: Glucose42; Other: Oral Glucose Tolerance Test

INTERVENTIONS:
Other: Glucose100
  Arms: Glucose100
Other: Glucose50
  Arms: Glucose50
Other: Glucose42
  Arms: Glucose42
Other: Oral Glucose Tolerance Test — For each OGTT, subjects will consume 50g of sweetener dissolved in water at a comfortable pace within 10 minutes. Blood samples for plasma glucose and insulin will be taken at -20, 0, 15, 30, 45, 60, 90 and 120 min after consuming the glucose drink. Plasma fructose will be tested at baseline, 30, 60, 90 and 120 minutes.
  Other Names: OGTT

SUMMARY:
The purpose of this study is to determine the glycemic index of commonly consumed sweeteners.

DETAILED DESCRIPTION:
This three arm study is intended to add to scientific knowledge by providing accurate assessments of the glycemic index commonly consumed food items. This will be used in the scientific literature to assess the glycemic index of foods containing various sweeteners. Participants will be monitored for a total of 10 weeks.

The glycemic index is defined as the "incremental area under the glucose response curve after standard amount of carbohydrate relative to that of a control food (white bread or glucose) is consumed." In general, the glycemic index quantifies the relative effect of the carbohydrate content of the food on resultant blood glucose.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-24.9 (lean)
* no medications
* no weight changes over the previous 6 months (defined as >=10% change in body weight)

Exclusion Criteria:

* current active participation in a weight loss program (dietary or physical activity focused)
* prior bariatric surgery
* significant medical condition such as cardiac or pulmonary disease, coagulopathy, gastrointestinal disorder, or known history of Type 1 or Type 2 diabetes
* women who are pregnant or lactating
* medications (except for oral contraceptives, thyroxins, drugs for hypertension, drugs for osteoporosis, or vitamins and minerals)
* no major medical or surgical event requiring hospitalization in the past 3 months
* no disease or drugs that influence digestion

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-10; Primary Completion 2017-12 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Mean Glycemic Index | 2 hours
  The mean glycemic index of participants will be calculated by averaging the 3 calculated glycemic index values for each of the 3 types of sweetener. Each participant will be randomly given 1 of 3 the commonly consumed sweeteners three different times over a nine week period- for a total of 3 observations per arm.
  Glycemic index is measured by giving test subjects the commonly consumed sweetener, and then measuring blood glucose response over a two hour time period using an Oral Glucose Tolerance Test. That response is then compared against a reference (glucose) and averaged across all subjects to get a relative index value.
  The glycemic index (GI) is a ranking of carbohydrates on a scale from 0 to 100 according to the extent to which they raise blood sugar levels after eating. (http://www.glycemicindex.com/about.php)

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Baseline
  BMI will be captured at the baseline visit, it will calculated using the formula Weight in Kilograms / ( Height in Meters x Height in Meters)
Body Mass Index (BMI) | 9 weeks
  BMI will be captured at the 9 weeks visit, it will calculated using the formula Weight in Kilograms / ( Height in Meters x Height in Meters)
Percent Fat Mass | Baseline
  Percent fat mass at baseline will be captured using the Tanita Body Fat Analyzer.
Percent Fat Mass | 9 weeks
  Percent fat mass at 9 weeks will be captured using the Tanita Body Fat Analyzer.
Total Fat Mass | Baseline
  Total fat mass at baseline will be captured using the Tanita Body Fat Analyzer.
Total Fat Mass | 9 weeks
  Total fat mass at 9 weeks will be captured using the Tanita Body Fat Analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Shapiro, MD, Principal Investigator — Yale University; Ania M Jastreboff, MD, PhD, Principal Investigator — Yale University; Robert S Sherwin, MD, Principal Investigator — Yale University
Locations (1):
- Yale Center for Clinical Investigation Church Street Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ludwig DS. The glycemic index: physiological mechanisms relating to obesity, diabetes, and cardiovascular disease. JAMA. 2002 May 8;287(18):2414-23. doi: 10.1001/jama.287.18.2414. PMID 11988062